CLINICAL TRIAL: NCT00390533
Title: An Eight-Week, Multicenter, Randomized, Double-blind, Placebo-controlled Study, to Evaluate the Efficacy, Safety and Tolerability of Two Fixed Doses (100 and 30 mg Once Daily) of Saredutant in Patients With Generalized Anxiety Disorder
Brief Title: An Eight-week Study to Evaluate the Efficacy and Safety of 2 Doses of Saredutant in Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5582; SR48968
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Generalized Anxiety
Keywords: Anxiety; clinical trials
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — SR 48968

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saredutant 30 mg (Experimental): Saredutant 30 mg once daily for a maximum of 8 weeks
  Interventions: Drug: Saredutant
- Saredutant 100 mg (Experimental): Saredutant 100 mg once daily for a maximum of 8 weeks
  Interventions: Drug: Saredutant
- Placebo (Placebo Comparator): Placebo for saredutant once daily for one week during the screening phase and for a maximum of 8 weeks during the acute phase
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saredutant — oral administration (capsules)
  Arms: Saredutant 100 mg; Saredutant 30 mg
Drug: Placebo — oral administration (capsules)
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the efficacy of two fixed doses (100 mg and 30 mg once daily) of saredutant compared to placebo in patients with generalized anxiety disorder. The secondary objectives are to evaluate the efficacy of saredutant on disability and quality of life in patients with generalized anxiety disorder, and to evaluate blood levels of saredutant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized anxiety disorder as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria and confirmed by the Mini International Neuropsychiatric Interview (MINI) Plus Generalized Anxiety Disorder module.

Exclusion Criteria:

* Total score of less than 22 on the HAM-A.
* Montgomery-Asberg Depression Rating Scale (MADRS) total score greater than 18.
* Patients with a current history (within 6 months) of major depressive disorder or history or presence of bipolar disorders or psychotic disorders.
* Patients with alcohol dependence or abuse or substance dependence or abuse in the past 12 months except nicotine or caffeine dependence.
* Patients who have used the following prior to entry into Acute Phase: antipsychotics within 3 months, antidepressants including Monoamine Oxidase Inhibitors (MAOIs) within 1 month, anxiolytics within 2 weeks, mood-stabilizer (lithium, anticonvulsants) within 1 month, and/or high dose or prolonged benzodiazepine (continuous use for 3 months prior to admission) use.

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 56 of treatment in the Hamilton Anxiety Rating Scale (HAM-A) total score. | 56 days

SECONDARY OUTCOMES:
Change from baseline to Day 56 of treatment in the Clinical Global Impression Severity of Illness score. | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia